CLINICAL TRIAL: NCT01731613
Title: Adjustable Fortification of Human Milk Fed to Chinese Preterm Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Collaborators: Mead Johnson Nutrition (Industry)
Responsible Party: Principal Investigator, Danhua Wang, Professor, Peking Union Medical College Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 8648
Record Dates: First submitted 2012-11-05; First posted 2012-11-22 (Estimated); Last update posted 2017-11-28 (Actual); Status verified 2017-11

CONDITIONS: Infant, Premature, Diseases
MeSH Terms: conditions — Infant, Premature, Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard Fortification (Active Comparator): receive human milk fortified with human milk fortifier(HMF) in the standard amount (4 packs /100 ml of HM) throughout the study
  Interventions: Dietary Supplement: human milk fortifier
- Adjustable fortification (Experimental): encompasses increasing/decreasing the amount of human milk fortifier(HMF) and adding supplemental protein guided by periodic determinations of the protein concentration of human milk (PCHM), body weight, blood urea nitrogen(BUN)
  Interventions: Dietary Supplement: human milk fortifier

INTERVENTIONS:
Dietary Supplement: human milk fortifier — Then fortification with human milk fortifier will be initiated at different levels according to the body weight of infants, the protein concentration of human milk and blood urea nitrogen
  Other Names: HMF

SUMMARY:
This clinical trial will compare how the individualized and fortified human milk feeding will help a premature infant grow.

DETAILED DESCRIPTION:
A total of 60 premature infants who will be randomized to receive either a standard fortification regimen (n=30) or an adjustable fortification regimen (n=30). The adjustable fortification regimen encompasses increasing / decreasing the amount of fortifier and adding supplemental protein guided by periodic determinations of the protein concentration in human milk (PCHM), body weight and blood urea nitrogen (BUN). Growth rate, tolerance of enteral feeding, days to achieve 100kcal/kg/d through enteral feeding, length of parenteral nutrition and NICU stays will be measured and compared between groups.

ELIGIBILITY:
Inclusion Criteria:

* Less than 34 weeks gestational age at birth
* Birth weight within 800-1800 grams
* Exclusively or mostly breastfed (greater than 80% if the feeding volume)
* Tolerated enteral feedings of 60 ml/kg/d
* Remain in the Neonatal Intensive Care Unit at least 14 days prior to hospital discharge,remain in the Neonatal Intensive Care Unit at least 10 days after enrollment
* Signed Informed Consent

Exclusion Criteria:

* Small for gestational age
* Infants currently receiving ventilation therapy
* Major congenital malformations
* Suspected or documented systemic or congenital infections
* Evidence of cardiac, respiratory, endocrinologic, hematologic, gastrointestinal, or other systemic diseases that may impact growth
* Severe intraventricular hemorrhage (greater than grade II) or periventricular leukomalacia
* Suspected or documented maternal substance abuse
* Infants currently receiving glucocorticoids or infants who have received glucocorticoids within the past 28 days

Ages: 10 Days to 40 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 51 (Actual)
Dates: Start 2012-08 (Actual); Primary Completion 2017-08 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Time to reach 100kcal/kg/d of enteral nutrition | participants will be followed until discharge, an expected average of 2 weeks
  Days to reach 100kcal/kg/d of enteral nutrition
The weight gain velocity during hospitalization | participants will be followed until discharge, an expected average of 2 weeks
  The weight gain velocity(g/kg/d)

SECONDARY OUTCOMES:
The protein and energy ratio of enteral nutrition each week after enrollment | participants will be followed until discharge, an expected average of 2 weeks
  The protein and energy ratio(g/100kcal)
Time to reach 2000g of body weight | participants will be followed until discharge, an expected average of 2 weeks
  Days to reach 2000g of body weight
metabolic indicators after enrollment, including BUN,prealbumin, albumin | participants will be followed until discharge, an expected average of 2 weeks
  BUN(mmol/L), prealbumin(mg/L), albumin(g/L)

CONTACTS AND LOCATIONS:
Overall Officials: Danhua Wang, Professor, Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No